CLINICAL TRIAL: NCT03394690
Title: the Evaluation of Green Coffee Extract Supplementation on Leptin, Ghrelin, Adiponectin,Anthropometric Measurements, Lipid Profile in Breast Cancer Survivors
Brief Title: Effects of Green Coffee Extract Supplementation on Leptin, Ghrelin, Adiponectin,Anthropometric Measurements, Lipid Profile in Breast Cancer Survivors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Nutrition and Food Technology Institute (Other)
Responsible Party: Principal Investigator, Dr Azita Hekmatdoost, Principal Investigator, National Nutrition and Food Technology Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 911
Record Dates: First submitted 2017-12-26; First posted 2018-01-09 (Actual); Last update posted 2018-01-09 (Actual); Status verified 2017-12

CONDITIONS: Breast Cancer Survivors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- green coffe (Active Comparator): green coffe 2 capsuls of green coffe
  Interventions: Dietary Supplement: green coffee
- control (Placebo Comparator): 2 capsuls of placebo
  Interventions: Other: control

INTERVENTIONS:
Dietary Supplement: green coffee — 2 capsuls
  Arms: green coffe
Other: control — 2 capsuls
  Arms: control

SUMMARY:
To study the effects of green coffee supplement on leptin, adiponectin, ghrelin, anthropometric measurements, lipid profile in breast cancer survivors.50 breast cancer survivors who their treatment is over and referred to follow breast cancer clinic with will be randomly allocated to receive placebos or 2 capsules green coffe for 12 weeks; both groups will be advised to adherence the investigators' diet and exercise program too. At the first and the end of the intervention, leptin, adiponectin, ghrelin, anthropometric measurements, lipid profile will be assessed and compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 to 70 years
* Body Mass Index (BMI) between 25-40 treatment is over

Exclusion Criteria:

* -Taking any kind of supplement for weight reduction
* pregnancy or lactation
* Professional athletes

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-03-12 (Estimated); Primary Completion 2019-02-12 (Estimated); Study Completion 2019-08-12 (Estimated)

PRIMARY OUTCOMES:
gherlin | 12 weeks
  assed by elisa
Adiponectin | 12 weeks
  assed by elisa
Leptin | 12 weeks
  assed by elisa

SECONDARY OUTCOMES:
body mass index | 12 weeks
  The body mass index (BMI) or Quetelet index is a value derived from the mass (weight)

CONTACTS AND LOCATIONS:
Locations (1):
- National Nutrition and Food Technology Research Institute, Tehran, Iran